CLINICAL TRIAL: NCT04730908
Title: Dentifrice With Innovative Remineralizing Technology
Acronym: REFIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Fabio Correia Sampaio, Professor, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: REFIX-UFPB
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Initial Dental Caries
Keywords: caries, white spot lesions, fluoride
MeSH Terms: interventions — Dentifrices; Toothpastes

STUDY DESIGN:
Intervention Model Description: Crossover study testing 4 dental gel for brushing teeth. the brushing period of use :7 days, 3 times daily with wahs-out periods of one week.
Who Masked: Participant, Care Provider, Investigator
Masking Description: the products are coded with different color in the label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- G0 - placebo (Placebo Comparator): Dental gel without fluoride in the composition
  Interventions: Other: DENTIFRICE
- G1: Daily Regenerator Dentalclean Neutro (RDCN) (Sham Comparator): 1450 ppm F- of sodium fluoride and tetrasodium pyrophosphate (Refix technology). NEUTRAL pH
  Interventions: Other: DENTIFRICE
- G2: Sensodyne Repair & Protect (SRP) (Active Comparator): 1426 ppm of sodium fluoride and calcium sodium phosphosilicate 5% (NOVAMIN technology).
  Interventions: Other: DENTIFRICE
- G3: Daily Regenerator Dentalclean Acid (RDCA) (Experimental): 1450 ppm F- of sodium fluoride and tetrasodium pyrophosphate (Refix technology). ACIDIC FORMULA
  Interventions: Other: DENTIFRICE
- G4: Colgate Total Daily Repair (CTDR) (Active Comparator): 1450 ppm F- of as sodium fluoride, 0.30% triclosan, arginine, tetrasodium pyrophosphate.
  Interventions: Other: DENTIFRICE

INTERVENTIONS:
Other: DENTIFRICE — GEL -DENTIFRICE FOR BRUSHING TEETH
  Other Names: TOOTHPASTE

SUMMARY:
Objective: The aim of this study is to evaluate in vivo dentifrices containing different active ingredients in fluoride (F) retention in saliva and dental biofilm. Material and methods: The dentifrices used in the study were: G1- Daily Regenerator Dentalclean Neutral (RDCN); G2- Sensodyne Repair & Protect (SRP); G3- Daily Regenerator Dentalclean Acid (RDCA), G4- Colgate Total Daily Repairc (CTDR). A double-blind, randomized crossover clinical study was conducted with eighteen residents of a city without a water fluoridation program. Biofilm and saliva samples were collected 1h and 12h after the last brushing for biofilm and, 1 to 60 minutes and 12 hours for saliva. The concentrations of F in saliva and biofilm were analyzed by specific electrode using the hexamethyldisiloxane facilitated diffusion technique (HMDS). Data were analyzed by repeated measures ANOVA followed by the Bonferroni test (p <0.05). Area under the curve (AUC) was calculated for saliva data. Result: No significant difference was observed between the groups regarding the retention of F in saliva. However, the largest area under the curve values in saliva were found for groups G3 and G4. The highest median values of F-biofilm were found in G3 for 1h and 12h collection times. Conclusion: The toothpaste containing Refix (RDCA) technology presented the most promising results for fluoride retention in oral exposure biomarkers.

DETAILED DESCRIPTION:
A randomized, duple-blind crossover clinical trial study was performed to evaluate the bioavailability of intraoral fluoride in biomarkers of exposure (biofilm and saliva) after the use of dentifrice with experimental fluoride for one week, with wash-out periods between them. The biofilm was collected 1 hour (h) and 12h after toothbrushing, and saliva was collected 1h (T1, T15, T30, T45, T60 min) and 12h. The data was obtained by potentiometry (ion selective electrode) for fluoride in these samples.

Study population The sample size was determined by sample calculation [25], according to previous studies [26], α = 5%, β = 10%, and a dropout ratio of 10%. Eighteen individuals with an average of 26 years old, including both males and females, participated in this study. The eligibility criteria were people over 18 years old, without systemic commitment and living in the city of João Pessoa-Paraíba, without water fluoridation (< 0.1 μg/mL F). Individuals were excluded if they used drugs that interfere with biofilm formation and salivary flow or fluoride products (> 5000 ppm) in the last 4 weeks, used orthodontic appliances, or had cavity lesions, periodontal disease, and/or tooth sensitivity.

Experimental Dentifrices The participants were allocated randomly to use the following experimental dentifrices according to table 1. They were coded by an independent investigator not involved in the trial. A simple randomization was performed taking into account a cross design. The unit of randomization was "dentifrice", so all dentifrices had the same chance of being selected. The design of the study was created for each participant and for each new one another draw was made.

Clinical Stage First, the participants were submitted to dental prophylaxis and scraping to remove all biofilm and dental calculus. They used a placebo, dentifrice without fluoride, for 7 days. Then, the Whitford protocol was followed [16]. Briefly, the subjects were instructed to brush their teeth three times/day for 1 min (transversal technique) and also to rinse their mouths after brushing with 10 mL of water. On the seventh day, the subjects were instructed to brush only the occlusal surfaces and do not use dental floss, to allow biofilm accumulation. After going to bed, they abstained from eating or drinking anything except water and did not brush their teeth. The next morning, after 12 hours of last brushing, and fasting, the first samples of saliva and biofilm (upper and lower right hemi-arch) were collected. Then, the volunteers brushed the occlusal surfaces for 1 min. Soon after, saliva samples were collected in the following times: t1, t15, t30, t45, and t60 minutes. Biofilme samples (left side) were collected later (1 hour after brushing). Resting saliva was collected for 5 minutes. The biofilm was collected from all tooth surfaces, in both buccal and lingual areas, using a 3S hollenback spatula, from which the samples were immediately transferred to an eppendorff tube, centrifuged and subsequently dried at 90°C for two hours and then weighed. The saliva samples were centrifuged at 6,000 rpm for 10 minutes in order to separate the saliva debris.

Determination of the concentration of fluoride The samples were analyzed by the hexamethyldisiloxane (HMDS) facilitated diffusion method of Taves [20] modified by Whitford [21]. The analyzes were performed with a fluoride specific electrode (model 9409; Orion Research) and a potentiometer (model EA 940; Orion Research, Cambridge, MA, USA) (Model 720 A Orion). Fluoride standards (1-100 nM) were used to prepare calibration curves.

Statistical analysis The data were analyzed using descriptive and inferential statistics, using the statistical program SPSS - v. 21.0 and software Graphpad. The Shapiro-Wilk test was applied to test the normality of the in vivo study data (n <50). Nonparametric tests were performed. The area under the curve (AUC) was calculated by taking baseline values (12 h after the last brush) up to 60 min after the last brush to indicate the effectiveness of F retention in saliva over time. For the purpose of comparing the concentration of F in saliva and biofilm between the groups, the ANOVA test of repeated measures was performed followed by the Bonferroni post-test. The relationship between the concentrations of biofilm and salivary fluoride was determined using Spearman's correlation coefficient. This study assumed a significance level of 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria were people over 18 years old, without systemic commitment and living in the city of João Pessoa-Paraíba, without water fluoridation (< 0.1 μg/mL F).

Exclusion Criteria:

* Individuals were excluded if they used drugs that interfere with biofilm formation and salivary flow or fluoride products (> 5000 ppm) in the last 4 weeks, used orthodontic appliances, or had cavity lesions, periodontal disease, and/or tooth sensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-02-12 (Estimated); Study Completion 2023-04-12 (Estimated)

PRIMARY OUTCOMES:
FLUORIDE IN SALIVA | 12 hours
  Concentration of fluoride in saliva after brushing teeth
FLUORIDE IN DENTAL PLAQUE | 12 hours
  Concentration of fluoride in dental biofilm after brushing teeth

CONTACTS AND LOCATIONS:
Overall Officials: FABIO SAMPAIO, PhD, Principal Investigator — Universidade Federal da Paraíba
Locations (1):
- Federal University of Paraíba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No